CLINICAL TRIAL: NCT04754204
Title: Mobile Cardiac Telemetry and Advanced Multi-Parameter Monitoring in Patients Wearing a Novel Device
Brief Title: Mobile Cardiac Telemetry and Advanced Multi-Parameter Monitoring in Patients
Acronym: MAPS
Status: Completed | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0234
Record Dates: First submitted 2021-02-09; First posted 2021-02-15 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Arrhythmia
Keywords: cardiac; arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients indicated for Mobile Cardiac Telemetry Monitoring: Patients indicated for Mobile Cardiac Telemetry Monitoring while meeting inclusion/exclusion criteria and enrolled in sequential manner.
  Interventions: Device: Arrhythmia Management System (AMS)

INTERVENTIONS:
Device: Arrhythmia Management System (AMS) — AMS records rhythm, heart rate, subject-reported symptoms, and multiple parameters that include respiration rate, activity and body posture.

SUMMARY:
To determine the associations among biometric data, arrhythmias, subject-reported symptoms and subject wellness.

DETAILED DESCRIPTION:
The Arrhythmia Management System records rhythm, heart rate, subject-reported symptoms and multiple parameters that include respiration rate, activity and body posture. These biometric data could provide clinicians better insight into the context of the detected arrhythmias, subject-reported symptoms and wellness status. Hence, the purpose of the study to determine the associations among biometric data, arrhythmias, symptoms and subject wellness.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who require monitoring for non-lethal cardiac arrhythmias
* Subjects who have an indication for mobile cardiac telemetry (MCT) monitoring
* Subjects 21 years of age or older

Exclusion Criteria:

* Subjects with an implantable cardiac device such as left ventricular assistive device, pacemaker, implanted cardioverter defibrillator (ICD), cardiac resynchronization therapy device, subcutaneous ICD's, pressure monitors and loop monitors
* Subjects with wearable cardioverter defibrillator, Holter monitors, wearable event recorders, and other mobile cardiac telemetry devices at the same time
* Subjects currently hospitalized
* Subjects with a skin condition preventing them from wearing the AMS device
* Subjects who are non-ambulatory
* Subjects who are self-reporting to be pregnant
* Subjects participating in another study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects, 21 years or older who:
  1. Require mobile cardiac telemetry monitoring for the detection of non-lethal cardiac arrhythmias
  2. Are without any cardiac implantable electronic devices, including loop recorders
  3. Are without wearable cardioverter defibrillator
  4. Are without Holter monitors, wearable event recorders, and other mobile cardiac telemetry devices at the same time
  5. Are not currently hospitalized
  6. Do not have any skin condition that would prevent them from wearing the AMS device
  7. Are not non-ambulatory
  8. Are not reporting to be pregnant
  9. Are not participating in another clinical study
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Biometric Data Associations to Arrhythmias | 30 days
  MCT Data Sets
Biometric Data Associations to Subject-Reported Symptoms | 30 days
  MCT Data Sets
Biometric Data Associations to Subject Wellness | 30 days
  MCT Data Sets

SECONDARY OUTCOMES:
Clinician Use of Biometric Data Associations to Arrhythmias | 30 days
  Clinical Case Report Forms
Clinician Use of Biometric Data Associations to Subject-Reported Symptoms | 30 days
  Clinical Case Report Forms
Clinician Use of Biometric Data Associations to Wellness Status of Subject | 30 days
  Clinical Case Report Forms

CONTACTS AND LOCATIONS:
Overall Officials: Ramu Perumal, PhD, Study Chair — Zoll Services LLC
Locations (20):
- United States (20):
  - Comprehensive Cardiovascular Medical Group, Bakersfield, California
  - Cardiovascular Innovation and Research Center, Long Beach, California
  - Heartbeat Cardiovascular Medical Group, Los Angeles, California
  - Interventional Cardiology Group, West Hills, California
  - Flagler Hospital/Flagler Health, Jacksonville, Florida
  - Cardiovascular Institute of Central Florida, Ocala, Florida
  - First Coast Heart and Vascular Center, Saint Augustine, Florida
  - Cardiovascular Research of Northwest Indiana, Munster, Indiana
  - Cardiovascular Research of Northwest, Munster, Indiana
  - Jackson Heart Clinic, Jackson, Mississippi
  - Trinity Medical, Cheektowaga, New York
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Erlanger Health System, Chattanooga, Tennessee
  - ClinicalTex Research LLC d/b/a PharmaTex Research, Amarillo, Texas
  - Texas Cardiology Associates of Houston, Kingwood, Texas
  - Heart Rhythm Specialists, McKinney, Texas
  - CardioVoyage, McKinney, Texas
  - Orion Medical Research, Pasadena, Texas
  - Daniel W. Gottlieb, MD, PS, Burien, Washington
  - St. Mary's Medical Center, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No